CLINICAL TRIAL: NCT06915025
Title: A Randomized Phase 3 Trial Evaluating the Safety & Efficacy of IP IMNN-001 Administered in Combination w/ Standard Neoadjuvant & Adjuvant Chemotherapy in Newly Diagnosed Patients w/ Advanced EOC, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Phase 3 Trial Evaluating the Safety & Efficacy of IMNN-001 Administered in Combination w/ Standard NACT & Adjuvant Chemotherapy in Newly Diagnosed Patients w/ Advanced EOC, Fallopian Tube or Primary Peritoneal Cancer
Acronym: OVATION-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Imunon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201-24-301
Record Dates: First submitted 2025-04-01; First posted 2025-04-07 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Epithelial Ovarian Cancer; Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: IMNN-001; GEN-1; OVATION-3
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — GEN-1; Paclitaxel; Carboplatin; olaparib; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm: IMNN-001 + SOC Chemotherapy + SOC Maintenance Therapy (Experimental): IMNN-001 in combination with standard neoadjuvant and adjuvant chemotherapy followed by standard of care maintenance therapy
  Interventions: Drug: IMNN-001 (IL-12 Plasmid Formulated with PEG-PEI-Cholesterol Lipopolymer); Drug: Paclitaxel; Drug: Carboplatin; Drug: Olaparib; Drug: Niraparib
- Control Arm: SOC Chemotherapy + SOC Maintenance Therapy (Active Comparator): Standard neoadjuvant and adjuvant chemotherapy followed by standard of care maintenance therapy.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Olaparib; Drug: Niraparib

INTERVENTIONS:
Drug: IMNN-001 (IL-12 Plasmid Formulated with PEG-PEI-Cholesterol Lipopolymer) — 100 mg/m2 IP given weekly during frontline treatment
  Other Names: GEN-1
  Arms: Experimental Arm: IMNN-001 + SOC Chemotherapy + SOC Maintenance Therapy
Drug: Paclitaxel — 175 mg/m2 IV given every 21 days for 6 cycles during frontline treatment
Drug: Carboplatin — AUC 6 IV given every 21 days for 6 cycles during frontline treatment
Drug: Olaparib — Olaparib (300 mg orally every 12 hours for 2 years) for patients with somatic or germline BRCAmut.
  Other Names: Lynparza
Drug: Niraparib — Niraparib (200-300 mg orally daily for 3 years; dosing based on participant's weight and platelet counts) for either HRD/BRCAmut & HRD/BRCAwt.
  Other Names: Zejula

SUMMARY:
This is a randomized, adaptive, open label, multicenter trial to evaluate the safety and efficacy of intraperitoneal (IP) IMNN-001 plus chemotherapy compared to chemotherapy alone.

DETAILED DESCRIPTION:
Eligible participants will be randomly assigned 1:1 to receive either chemotherapy plus IMNN-001 or chemotherapy alone, followed by standard of care maintenance therapy.

Randomization will stratify by confirmed biomarker tumor homologous recombination deficiency status and stage of cancer.

On both arms, the chemotherapy regimen will consist of paclitaxel 175 mg/m2 IV over 3 hours followed by carboplatin AUC 6 IV over 1 hour on Day 1 of each cycle. This will be repeated every 3 weeks for a total of 6 cycles, 3 in the neoadjuvant period and 3 in the adjuvant period following interval debulking surgery (IDS). On the experimental arm, IMNN-001 at a dose of 100 mg/m2 will be administered IP on Days 8 and 15 of the first chemotherapy cycle and then on Days 1, 8, and 15 of all subsequent 5 chemotherapy cycles for a total of 17 treatments in the neoadjuvant and adjuvant settings. When given on the same day as chemotherapy, IMNN-001 should be given at least 30 minutes after completion of carboplatin infusion. IDS will take place after 3 cycles of neoadjuvant chemotherapy (NACT) + IMNN-001 for 8 doses. Additional cycles of NACT are allowed at the discretion of the investigator but with discussion with the medical monitor.

An independent Data Monitoring Committee (iDMC) will monitor participants' safety and study conduct throughout the course of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be female, ≥18 years of age, able to understand the study procedures, and agree to participate in the study by providing written informed consent.
2. Participants with a histologically confirmed diagnosis of high-grade non-mucinous epithelial ovarian (serous, endometrioid, carcinosarcoma, mixed epithelial pathologies), fallopian tube or peritoneal cancer that is Stage IIIB/C or IV according to the International Federation of Gynecology and Obstetrics (FIGO) or tumor, node and metastasis staging criteria.
3. Participants eligible to receive neoadjuvant chemotherapy.
4. Participants will provide a tumor tissue sample at pre-screening or screening, via laparoscopy or image guided core biopsy for determination of confirmed biomarker tumor status (HRD vs. HRP). See biomarker status definitions in the section below.
5. Participants of childbearing potential must have a negative serum pregnancy test (beta human chorionic gonadotropin) within 14 days prior to initiation of protocol therapy and be practicing an effective form of contraception. If applicable, participants must discontinue breastfeeding prior to study entry.
6. Participants must have adequate:

   1. Bone marrow function: Absolute neutrophil count (ANC) greater than or equal to 1,500/µl. Exceptions may be made in patients with benign ethnic neutropenia >800/ul with approval of a medical monitor. This ANC cannot have been induced or supported by granulocyte colony stimulating factors. Platelets greater than or equal to 100,000/µl.
   2. Renal function: eGFR > 60 ml/min/1.73m2
   3. Hepatic function: Bilirubin ≤ 1.5 x ULN. SGOT (AST) and SGPT (ALT) ≤ 3.0 x ULN and alkaline phosphatase ≤ 2.5 x ULN. Exceptions due to hepatic metastases can be considered in consultation with medical monitor.
   4. Neurologic function: Neuropathy (sensory and motor) less than or equal to Grade 1 as defined by CTCAE version 5.0.
7. Participants must have an ECOG score of 0, 1 or 2.
8. Participants should be free of active infection requiring parenteral antibiotics or a serious uncontrolled medical illness or disorder within 4 weeks of study entry.
9. Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to the first treatment. Continuation of hormone replacement therapy is permitted.

Exclusion Criteria:

1. Participant who has received prior treatment with IMNN-001.
2. Participant who has received oral or parenteral corticosteroids (>10 mg prednisone) within 2 weeks of first dose of IMNN-001 (if applicable) or who have a clinical requirement for ongoing systemic immunosuppressive therapy such as chronic steroid use not related to chemotherapy administration.
3. Participant has mucinous, germ cell, transitional cell, clear cell, undifferentiated, or non-epithelial ovarian cancer.
4. Participant has low-grade or Grade 1 epithelial ovarian cancer.
5. Participant of childbearing potential, not practicing adequate contraception, participant who is pregnant, or participant who is breastfeeding are not eligible for this trial.
6. Participant has a bowel obstruction by clinical symptoms or computed tomography (CT) scan, sub-occlusive mesenteric disease, abdominal or gastrointestinal fistula, gastrointestinal perforation, or intra-abdominal abscess.
7. Participant has been diagnosed and/or treated with any therapy for invasive cancer <3 years from study enrollment, completed adjuvant chemotherapy and/or targeted therapy at least 3 years from enrollment, or completed adjuvant hormonal therapy less than 4 weeks from enrollment.
8. Participant with definitively treated non-invasive malignancies such as cervical carcinoma in situ, ductal carcinoma in situ, grade 1 or 2 Stage IA endometrioid endometrial cancer, or non-melanomatous skin cancer are allowed.
9. Participant with concurrent severe medical problems unrelated to the malignancy that would significantly limit full compliance with the study or expose the participant to extreme risk or decreased life expectancy.
10. Participant has known active hepatitis or HIV with detectable viral load.
11. Participant has a known contraindication or uncontrolled hypersensitivity to the components of paclitaxel, carboplatin, IMNN-001, or their excipients.
12. Prior treatment for high-grade non-mucinous epithelial ovarian, fallopian tube, or peritoneal cancer (e.g., immunotherapy, anticancer therapy, surgery, radiation therapy).
13. Participant is receiving treatment for active autoimmune disease. "Active" refers to any condition currently requiring therapy. Examples of autoimmune disease include systemic lupus erythematosus, multiple sclerosis, inflammatory bowel disease and rheumatoid arthritis.
14. Participant who has received prior radiotherapy to any portion of the abdominal cavity or pelvis is excluded. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, if it was completed at least 3 years prior to registration, and the participant remains free of recurrent or metastatic disease.
15. Participant who has received prior chemotherapy for any abdominal or pelvic tumor is excluded. Participant may have received prior adjuvant chemotherapy for localized breast cancer, if it was completed at least three years prior to registration, and that the participant remains free of recurrent or metastatic disease.
16. Participant with history or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of treatment on this study.
17. Participant who will receive bevacizumab with the neoadjuvant or adjuvant treatment, or as maintenance will be excluded.
18. Participant with any condition/anomaly that would interfere with the appropriate placement of the IP catheter for study drug administration including abdominal surgery within 4 weeks of study entry (for reason other than IP port placement or laparoscopic diagnosis of epithelial ovarian cancer), intestinal dysfunction as defined in #6 above.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2032-10-31 (Estimated); Study Completion 2032-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 48 months
  Overall Survival is defined as the time (in months) from the date of randomization to the date of death by any cause.

SECONDARY OUTCOMES:
Chemotherapy Response Score | 12 weeks
  After the interval debulking surgery takes place, participants will be assessed for a chemotherapy response score by the pathologist and scored based on CRS3, CRS2, or CRS1.
Surgical Response | 12 weeks
  After the interval debulking surgery takes place, participants are scored in terms of their interval debulking status with a score of R0, R1, or R2.
Time to Second Line Treatment | 13 months
  Time to second line treatment is defined as the time (in months) from the date of randomization to the date of second line chemotherapy treatment or death, whichever occurs first.
Objective Response Rate | 12 weeks
  Objective Response Rate is defined as the proportion of participants with objective evidence of CR or PR prior to IDS. The evaluation of objective response rate will be based on investigator (site) assessment of the images following RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Premal H Thaker, M.D., Study Chair — Washington University School of Medicine
Locations (5):
- United States (5):
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Providence Cancer Institute, Portland, Oregon
  - Sanford Health, Sioux Falls, South Dakota
  - Erlanger Health, Chattanooga, Tennessee
  - Providence Sacred Heart Medical Center & Children's Hospital, Spokane, Washington